CLINICAL TRIAL: NCT00375661
Title: Phase 4 Study of Peg-interferon Plus Ribavirin Therapy for Prevention of Hepatocellular Carcinoma
Brief Title: Low-dose Peg-interferon Plus Ribavirin (IFN/RBV) for Prevention of Hepatocellular Carcinoma (HCC) Recurrence in Patients Who Had Surgery to Remove Primary HCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyoto University (Other)
Responsible Party: Principal Investigator, Hiroyuki Marusawa, Associate professor, Kyoto University
Organization: Kyoto University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: O2006-415
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatocellular carcinoma
MeSH Terms: conditions — Hepatitis C, Chronic; Carcinoma, Hepatocellular | interventions — Introns; Ribavirin

ARMS (1):
- interferon (No Intervention)
  Interventions: Drug: interferon-alfa-2b and ribavirin

INTERVENTIONS:
Drug: interferon-alfa-2b and ribavirin — Interferon, pnce per week plus daily ribavirin

SUMMARY:
The purpose of this study is to determine whether low-dose peg-interferon plus ribavirin therapy is effective in the prevention of hepatocellular carcinoma (HCC) in patients who had the curative resection of primary HCC.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Hepatocellular carcinoma due to Chronic Hepatitis C Virus Infection.
* Must be treated with curative treatment for primary tumor using either surgical resection or radiofrequency ablation therapy

Exclusion Criteria:

* No recurrence of hepatocellular carcinoma 3 months after the primary treatment
* Renal dysfunction

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-09; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse effect of interferon | During the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Chiba, M.D.,Ph.D., Study Chair — Kyoto University Hospital
Locations (2):
- Japan (2):
  - Department of Gastroenterology and Hepatology, Kyoto University Hospital, Kyoto
  - Osaka Red Cross Hospital, Osaka